CLINICAL TRIAL: NCT05121623
Title: Inappropriate Sexual Behaviour (ISB) of Patients Towards French General Practitioners: Prevalence, Nature and Impact on Professional Practice
Brief Title: Inappropriate Sexual Behaviour of Patients Towards French General Practitioners
Acronym: #MedTooFr
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/18
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Sex Behavior
MeSH Terms: conditions — Sexual Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Online auto-administered Questionnaire

SUMMARY:
Occupational sexual harassment (HS) has come to the fore in recent years, particularly with the #MeToo social movement that has encouraged women victims of sexual violence to speak out around the world. The medical profession is not exempt from this phenomenon, whether during the training or professional life of practitioners. In France, very little data is available on this subject, particularly among general practitioners. However, the specific nature of the doctor-patient relationship in general practice makes it a potentially high-risk setting. Furthermore, practitioners' experiences of inappropriate sexual behaviour (ISB) can lead to changes in professional practice, and can thus directly influence the quality of care provided to patients. It is also described in the literature that sexual harassment in physicians is independently associated with a decrease in job satisfaction and sense of security at work, and may be associated with an altered mental health status. To date, the only French studies on ISB and HS in medicine have focused on the period of medical study, and none have looked at the particular problem of the patient as perpetrator of the violence. It is in this context that it has been decided to set up this cross-sectional study with the aim of evaluating the prevalence of ISB occurring during consultations with French general practitioners, to describe their characteristics and to evaluate the responses provided and the repercussions on professional practice.

ELIGIBILITY:
Inclusion Criteria:

* Any general practitioner
* Male or female
* Sole or mixed private practice
* Installed or substitute
* Having completed their internship in general medicine
* With or without a thesis
* Practising alone, in a group practice or in a health centre -

Exclusion Criteria:

* Specialty other than general medicine
* Exclusive hospital or salaried activity
* Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: General practitioners in private practice in France.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Prevalence and nature of inappropriate sexual behaviour of patients towards general practitioners in private practice in France | Once at the inclusion visit
  Determined by auto-administered questionnaire (sociodemographic data, personal experience, author's characteristics, reactions and answers provided by the practitioners)

SECONDARY OUTCOMES:
Prevalence and nature of Inappropriate sexual behavior between men and women | Once at the inclusion visit
  To compare the prevalence and nature of Inappropriate sexual behavior according to the gender of the responding physicians determined by auto-administered questionnaire

OTHER OUTCOMES:
Risk factors associated with sexual inapropriate behavior | Once at the inclusion visit
  Identify the risk factors associated determined by auto-administered questionnaire (author's characteristics provided by the practitioners)
Responses of general practitioners to such a situation | Once at the inclusion visit
  Types of responses provided by general practitioners to such a situation determined by auto-administered questionnaire (answers provided by the practitioners)
Impact and changes on professional practice and personal life. | Once at the inclusion visit
  Describe the impact and changes on professional practice and personal life determined by auto-administered questionnaire (reactions provided by the practitioners)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No